CLINICAL TRIAL: NCT01740908
Title: Pilot Study for the Detection of Stem/Progenitor Cell Up-regulation Using Aldagen BRIGHT Technology in Peripheral Blood After Hyperbaric Oxygen Therapy (HBOT) Treatment
Brief Title: Stem Cell Quantification In Peripheral Blood After Hyperbaric Oxygen Therapy Treatments
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Restorix Research Institute, LLLP (Other)
Collaborators: Cytomedix (Industry); Island Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RRI-2012-05-STCELL-001; RF-STCELL-2012 (Other Grant/Funding Number: Restorix Foundation/Cytomedix)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Changes in Peripheral Blood Population Numbers and Type.
Keywords: hyperbaric oxygen; stem cell
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2C | interventions — Oxygen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hyperbaric Oxygen Treatment: Six healthy adult individuals (18-65 yrs), with no current, ongoing infection or chronic disease will be recruited for this study. Treatment study subjects will undergo a daily exposure to 2.0 ATA, 100% Oxygen for 90 minutes over 5 days.
  Interventions: Other: Hyperbaric Oxygen Treatment
- Baseline: Two healthy study subjects with no current, ongoing infection or chronic disease will be rectuited to serve as a baseline group. Study subjects will not be exposed to HBO, but will have blood drawn at the same time as the treatment group.

INTERVENTIONS:
Other: Hyperbaric Oxygen Treatment — Hyperabric oxygen will be delivered via a PerryPerry-Sigma Monoplace Hyperbaric Chambers. Oxygen is supplied by Air Gas, Seattle.
  All gases will meet Health Standards for oxygen and air. The hyperbaric chamber technicians employed by Restorix Health are trained health personnel who will be assisting our study participant and monitoring the HBO treatment. Oxygen will be delivered at a pressure of 2.0 ATA for 90 minutes, once a day for 5 consective days.
  Other Names: 100% Oxygen USP
  Groups: Hyperbaric Oxygen Treatment

SUMMARY:
This is an observational research study whose purposes are to see the effects of repeated hyperbaric oxygen therapy treatments on the levels of stem/progenitor cells in peripheral circulating blood following five days of treatment, 90 minutes per day at 2.0 atmospheres absolute in 100% USP Grade Oxygen. Hyperbaric oxygen has a greater oxygen concentration than air at sea level. In this research, the concentration of oxygen will be twice the level of oxygen at sea level.

ELIGIBILITY:
Inclusion Criteria:

Patients recruited will be healthy volunteers with no current, ongoing infection or chronic disease.

Exclusion Criteria:

We will exclude or delay the treatment if our patients have an active lung infection, develops cancer, if the patient cannot undergo pressurization/ depressurization because of eustachian-tube dysfunction and confinement anxiety. Any patient that cannot breathe without a respirator will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will reflect the racial and ethnic distribution that exists in the Anacortes metropolitan region.
  B- Skagit County, WA: White (91.4%), Black (0.9%), American Indian (2.6%), Asian or Pacific Islander (2.3%), Other (2.8%)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2012-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood analysis of circulating stem cells | 5 days
  Six treatment subjects and two control subjects will have two daily blood draws. Exposures of hyperabric oxygen (HBO) will occur daily over 5 consecutive days. The blood draws will occur prior to starting HBO exposure and after finishing with the HBO exposure. Control subjects will have their blood drawn at the same time as the treatment subjects, in ordert to establish a non-treatment baseline. The stem cell population that is resident in the peripheral blood will be analyzed using the cell sorting and cell identification system at Aldagen. Mononulcear cells will be gated on the basis of forward and side laser light scatter, and 250,000 events will be analyzed to determine the percentage of ALDHbr cells, and the expression of additional stem cell markers, such as CD45, CD34, and CD105.

CONTACTS AND LOCATIONS:
Locations (1):
- Restorix Wound Treatment Center at Island Hospital, Anacortes, Washington, United States

REFERENCES:
- [Background] Thom SR, Bhopale VM, Velazquez OC, Goldstein LJ, Thom LH, Buerk DG. Stem cell mobilization by hyperbaric oxygen. Am J Physiol Heart Circ Physiol. 2006 Apr;290(4):H1378-86. doi: 10.1152/ajpheart.00888.2005. Epub 2005 Nov 18. PMID 16299259